CLINICAL TRIAL: NCT04047524
Title: Trimodal Prehabilitation Programme Using Smart Watches and Mobile Applications in Patients Undergoing Major Abdominal Surgery: a Randomised Controlled Pilot Study
Brief Title: A Trimodal Prehabilitation Study for Patients Undergoing Major Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shira Baram (Other)
Collaborators: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Shira Baram, Research Project Manager, University of Manchester
Organization: University of Manchester (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 19_SURG_19
Record Dates: First submitted 2019-07-15; First posted 2019-08-06 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Pilot Study

STUDY DESIGN:
Intervention Model Description: Participants will be randomised sequentially i.e. 1:1 to receive either the Prehabilitation Programme or not
Masking Description: There is no masking. Both the investigator and participant will be aware of which arm they have been randomised to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation (Other): These participants will receive a home based prehabilitation programme for a period of 2-6 weeks prior to surgery and will be provided with a Fitbit Charge 2.
  Interventions: Other: Monitoring using a FitBit
- Control (Other): These participants will receive a Fitbit Flex and told to continue with their every day activity levels for a period of 2-6 weeks prior to surgery
  Interventions: Other: Monitoring using a FitBit

INTERVENTIONS:
Other: Monitoring using a FitBit — Each participant will receive a Fitbit. The Prehabilitaiton Group will receive a Fitbit Charge 2 and they will be able to review their progress on this and be required to increase their exercise activity and input information and data about the exercise they have completed each day during their participation in the study. The Control group will receive a Fitbit Flex and will not be required to review any of their activity or input any data and will be encouraged to continue with their daily activity rates i.e. not to change.

SUMMARY:
Prehabilitation programmes have the potential to reduce post-operative complications following abdominal cancer surgery by improving pre-operative fitness levels. Home-based prehabilitation programmes may be more cost effective than hospital-based programmes, but have issues with low compliance. The aims of our study are to assess whether mobile technologies such as smart watches and smartphone applications improve compliance with home-based prehabilitation programmes and to assess the effects of prehabilitation on pre-operative fitness levels in patients due to undergo major abdominal cancer surgery.

DETAILED DESCRIPTION:
30 patients due to undergo major abdominal cancer surgery at The Christie NHS Foundation Trust will be enrolled to a pilot randomised controlled trial. They will randomised to either a home-based trimodal prehabilitation programme, delivered by the use of FitBit Smart Watches and Smartphone applications, or a control group who will receive a FitBit for physical activity monitoring only, for a period of 2-6 weeks prior to surgery. The prehabilitation programme will include exercise, nutritional, and psychological components. Study outcomes will include 6MWT (6-minute walk test), HADS (hospital anxiety and depression score), steps per day, length of stay post-operatively, and post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

* be aged 18 years or over
* be able to consent to participate in the prehabilitation programme
* be undergoing major abdominal cancer surgery (including, but not limited to, cytoreductive surgery with hyperthermic intraperitoneal chemotherapy)
* have at least 2 weeks to their operation date
* be able to understand written and spoken English

Exclusion Criteria:

* patients have any health conditions which will prevent them from safely taking part in a home-based exercise programme. For example, but not limited to, patients who have recently (within the past 3 months) had a myocardial infarction or a stroke or patients who have end-stage renal disease but are not on dialysis. We will use the "Safety Reference Guide to support exercise services in people with cancer" in The Lancet published paper "Exercise as part of routine cancer care"(5) to aid the screening of patients suitability.
* they have any bone metastasis
* are already active users of a FitBit device

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2019-12-28 (Estimated); Study Completion 2019-12-28 (Estimated)

PRIMARY OUTCOMES:
Quantitative data collected via a Fitbit | Each participant will be monitored for a period of 2-6 weeks pre surgery
  Data will be collected to determine the number of participants whose physical activity increased and by how much during the study

SECONDARY OUTCOMES:
Qualitative data collected by questionnaire | Each participant will be monitored for a period of 2-6 weeks pre surgery
  Qualitative data will be collected from participants to identify their experience of the study
Quantitative data associated with participants weight at the start and end of the research intervention | Each participant will be monitored for a period of 2-6 weeks pre surgery
  Participants weight will be measured in kilograms at the start of their participation and then prior to surgery to determine if they were able to either maintain their weight or gain weight

CONTACTS AND LOCATIONS:
Overall Officials: Omer Aziz, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will not currently be shared with researchers outside of the study team

REFERENCES:
- [Derived] Waller E, Sutton P, Rahman S, Allen J, Saxton J, Aziz O. Prehabilitation with wearables versus standard of care before major abdominal cancer surgery: a randomised controlled pilot study (trial registration: NCT04047524). Surg Endosc. 2022 Feb;36(2):1008-1017. doi: 10.1007/s00464-021-08365-6. Epub 2021 Mar 15. PMID 33723969